CLINICAL TRIAL: NCT05644925
Title: Effects of Pressure-controlled Intermittent Coronary Sinus Occlusion (PiCSO) Therapy on miRNAs Expression and Absolute Microvascular Resistance by Continuous Thermodilution in ST-segment Elevation Myocardial Infarction (STEMI) Patients: PiCSO-STEMI TRIAL
Acronym: PiCSO-STEMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support for recruitment and follow-up activities.
Sponsor: Fundacio Privada Mon Clinic Barcelona (Other)
Collaborators: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PiCSO-STEMI
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anterior Myocardial Infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (1:1) to PiCSO group or standard PCI control group. Once randomized, PiCSO group patients will receive PiCSO therapy inside the catheterization laboratory.
Who Masked: Outcomes Assessor
Masking Description: The subjects as well as the investigator performing the procedure will not be blind to the study treatment. An independent experienced cardiologist, who will be blinded to all clinical data; will analyze anonymized Cardiac Magnetic Resonance (CMR) images for unbiased endpoints assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PICSO+PCI (Experimental)
  Interventions: Device: PiCSO Impulse System; Procedure: Percutaneous Coronary Intervention (PCI)
- Standard PCI (Active Comparator)
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)

INTERVENTIONS:
Device: PiCSO Impulse System — The PiCSO Impulse System is intended to reduce infarct size by intermittently occluding the coronary sinus outflow in patients undergoing a percutaneous coronary interventional procedure for myocardial infarction and presenting with Thrombolysis in myocardial infarction (TIMI) flow of 0 or 1.
  Arms: PICSO+PCI
Procedure: Percutaneous Coronary Intervention (PCI) — Minimally invasive procedures used to open clogged coronary arteries

SUMMARY:
In this study we pretend to determine the molecular (miRNAs expression, angiogenic and inflammatory biomarkers) and microcirculatory (assessed by the innovative continuous intracoronary thermodilution technique) effects of PiCSO compared to a standard PCI control group in patients with high-risk anterior STEMI. Then, we aim to assess the efficacy of these molecular biomarkers as prognostic tools. Also, we will evaluate the impact of PiCSO on the coronary microcirculation beyond the acute phase in the follow-up six months after STEMI. Finally, we will assess PiCSO influence on Heart Failure (HF) clinical variables and patients' quality of life including a cost-effectiveness assessment in the mid-term follow-up one year after the STEMI event.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Anterior STEMI (ECG with persistent elevation ≥ 2 mm (0.2 mV) in 2 or more contiguous anterior precordial leads (V2, V3, V4) in men or ≥ 1.5 mm (0.15 mV) in women.
3. Culprit lesion in proximal or mid Left Anterior Descending Artery (LAD).
4. Pre-PCI TIMI flow 0-1.
5. Symptoms consistent with myocardial ischemia (persistent chest pain, dyspnea, nauseas/vomiting, fatigue, palpitations or syncope) present for ≤ 12 hours.
6. The patient is eligible for primary PCI.
7. Informed consent received and signed for study enrollment.

Exclusion Criteria:

1. Contraindication to coronary angiogram or PCI.
2. Implants or foreign bodies in the coronary sinus.
3. Known allergies to polyurethanes, Polyethylene Terephthalate (PET) or stainless steel.
4. Known pregnancy or breastfeeding.
5. Known coagulopathy.
6. Known severe kidney disease (eGFR <=30 mL/min/1.73) and/or hemodialysis.
7. Known large pericardial effusion or cardiac tamponade.
8. Central hemodynamically relevant left-right shunt.
9. Previous MI or Coronary Artery Bypass Graft (CABG).
10. Previous history of stroke, transient ischemic attack (TIA) or reversible ischemic neurological deficit within last 6 months.
11. Cardiopulmonary resuscitated (CPR) cardiac arrest ≥ 5 minutes whom baseline neurologic status is not present.
12. Unconscious at presentation.
13. Need for circulatory support.
14. Need for invasive mechanical ventilation.
15. Need for temporal intravenous pacemaker.
16. Patient not suitable for femoral access.
17. Known contraindication for adenosine administration (severe asthma, complicated Atrioventricular (AV) block, critical aortic stenosis, severe cardiac arrhythmias, severe valve diseases).
18. Known epicardial stenosis greater than 50% distal to the culprit LAD lesion.
19. Active participation in another drug or device investigational trial.
20. Medical, social or psychological condition that limits the ability of patient to participate in the study.
21. Patients with definite or probable coronavirus disease 19 diagnosis within 2 weeks prior to STEMI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Superiority of PiCSO in reducing microvascular dysfunction | After primary PCI at time 0 after intervention
  To determine the superiority of PiCSO in reducing the microvascular dysfunction (defined as microvascular resistance >500 WU) as compared to standard of care

IPD SHARING:
Plan to Share IPD: No